CLINICAL TRIAL: NCT04519736
Title: Single Band (Alma) vs. Dual Band (Palomar) Pulsed Light Technology for the Treatment of Photodamage - a Split Face Comparison Study
Brief Title: Single Band vs. Dual Band Pulsed Light Technology for the Treatment of Photodamage - A Split Face Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALMA-500600-PL12DG
Record Dates: First submitted 2014-01-07; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2013-04

CONDITIONS: Photodamage
Keywords: Hyperpigmentation; Telangiectasias
MeSH Terms: conditions — Hyperpigmentation; Telangiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Harmony Dye-VL 500-600nm (Active Comparator): The left side of the face will be treated with the Single Band Alma Harmony Dye-VL 500-600nm device. Three treatments, administered in intervals of 21 +/- 2 days. Each full face treatment duration will be approximately 20-30 minutes .
  Interventions: Device: Single Band vs. Dual Band Pulsed Light Technology for the Treatment of Photodamage
- Palomar MaxG (Active Comparator): Right side of the face will be treated with the Dual Band Palomar MaxG device. Three treatments, administered in intervals of 21 +/- 2 days. Each full face treatment duration will be approximately 20-30 minutes .
  Interventions: Device: Single Band vs. Dual Band Pulsed Light Technology for the Treatment of Photodamage

INTERVENTIONS:
Device: Single Band vs. Dual Band Pulsed Light Technology for the Treatment of Photodamage

SUMMARY:
Both the Dye - VL 500 - 600 nm and the Dual band will improve significantly the appearance of Photo Damage with high efficacy including; safety, minimal discomfort and downtime.

ELIGIBILITY:
Inclusion Criteria:

The following are requirements for a potential subject's inclusion into the study:

* Male or female in good general health between 35 to 65 years of age.
* Must be willing to execute informed consent. Patient must also consent to having photos taken at each visit.
* A potential subject must exhibit:

Clinical diagnosis of photo damage affecting the face.

* For FEMALE PATIENTS OF CHILDBEARING POTENTIAL, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplanit®, Depo-Provena®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation.
* Must be willing to comply with study visits and complete the entire course of the study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from participation:

The following are exclusion criteria for subjects in this study:

* A subject that underwent a laser / light treatment on the face within 12 months, or any topical treatment on the face within 6 months.
* A subject with any UNCONTROLLED systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* A subject using any topical product containing a retinoid, retinol, or other vitamin A derivative within 3 months prior to or during the study period.
* A subject using any systemic steroid therapy within 6 months prior to or during the study period.
* A subject that has been treated with Botox/Dysport or filler/biostimulatory molecule injections to his/her face within the past 6 months.
* A subject using any topical medicated creams, lotions, powders, etc. on the treatment areas during the study period, other than the study treatment regimen within 14 days.
* A subject that has previously been treated with systemic retinoids within the past year (e.g., Accutane®, Roche Dermatologics).
* A subject with recently excessive facial exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing). During the study, when excessive sun exposure is unavoidable, subjects must wear appropriate protective clothing (e.g. hat, collar) and comply with the study dosing regimen of daily application of the dispersed sunblock.
* A subject with a recent history or active presence of any facial skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e. moderate to severe acne vulgaris, atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis, excessive facial hair or coloration).
* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, intrauterine device, abstinence, or spermicides and condoms used in combination)].
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.
* Subjects who are pregnant, breast-feeding, or planning a pregnancy. Females of childbearing potential, must be either:

  * using the same form (i.e. brand) and dosage regimen of an oral contraceptive pill or of a hormonal implant continuously for 3 months prior to study entry and continue during the entire study, or
  * willing to use a different form of birth control during the study other than any form of hormonal methods such as oral contraceptive pills and hormonal implants 30 day prior to study entry and during the entire study period. For the purpose of this study, the following are also considered acceptable methods of birth control: double-barrier methods (e.g.: condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control, should the subject become sexually active.

Ages: 35 Years to 60 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Photodamage | The investigator will evaluate the change in visual appearance of the treated area at 3 week, 6 week, 9 week treatments and before follow-up visit (3 months after the last treatment)
  Investigator Evaluation of Specific Signs of Photo Damage
  The investigator will evaluate the clinical improvement from the visual appearance of the treated area and from the fixed magnification clinical photographs according to the following Global Assessment scale (compared to baseline photographs):
  Global Aesthetic Improvement Scale (GAIS ) Rating Description
  1. = Very much improved 75%-99%
  2. = Much improved 50%-75% 3= Improved 25%-50% 4= No change 1%-25% 5=Worse <1%

SECONDARY OUTCOMES:
Photodamage | Investigator will evaluate the change in visual appearance of the treated area at 3 week, 6 week, 9 week treatments, and before follow up visit (three months after the last visit)
  Investigator Evaluation of Specific Signs of Photo Damage
  In addition, the Investigator will at each visit complete the Investigator Evaluation of Specific Signs of Photo Damage as seen below (for each of the handpieces):
  Poilikoderma of Civatte
  * None (0) = Normal
  * Trace (1) = Barely visible and localized
  * Mild (2) = Somewhat visible and diffuse
  * Moderate (3) = Visible and diffuse
  * Severe (4) = Extremely visible and dense
  Telangiectasias
  * None (0) = Normal
  * Trace (1) = Barely visible and localized
  * Mild (2) = Somewhat visible and diffuse
  * Moderate (3) = Visible and diffuse
  * Severe (4) = Extremely visible and dense
  Pigmented components of Photo Damage
  * None (0) = Normal
  * Trace (1) = Barely visible and localized
  * Mild (2) = Somewhat visible and diffuse

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Laser & Surgery Specialists of NY/NJ, Hackensack, New Jersey, United States